CLINICAL TRIAL: NCT00005679
Title: Pathobiological Determinants of Atherosclerosis in Youth (PDAY)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1049; R10HL033772 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Heart Diseases; Coronary Disease; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Heart Diseases; Coronary Disease; Coronary Artery Disease

SUMMARY:
To conduct a multicenter prevalence survey for characterizing pathologically the extent of atherosclerosis in the aortas and coronary arteries of young persons dying from accidental causes, suicide, or homicide.

DETAILED DESCRIPTION:
BACKGROUND:

The International Atherosclerosis Project (IAP) quantified atherosclerosis of the aorta and coronary arteries in over 31,000 persons age 10 to 69 who died between 1960 and 1965 in fifteen cities and countries throughout the world. The IAP established that the average severity of atherosclerosis differed widely in many parts of the world and that the differences correlated with mortality from ischemic heart disease. It also demonstrated that the fatty streaks of childhood were prevalent and severe in both boys and girls. Fibrous plaques generally first appeared between the ages of 20 and 30 and in proportion to the prevalence of ischemic disease in the adult population. Since the results of the IAP were first published in 1968, research into atherosclerosis has changed greatly from gross and microscopic morphological methods to manipulation of experimental animals, in vitro culture of arterial wall cells, and the application of micro-chemical, physical chemical, and immunological techniques to tissues.

The use of these newer techniques made it possible to test the hypothesis that a series of changes in the fatty streak between the ages of fifteen and twenty-five lead to the typical fibrous plaque and to test the hypothesis that lesions other than fatty streaks precede and may progress to fibrous plaques. The study also tested associations of the established risk factors for atherosclerosis with early stages of lesion progression as seen in young persons.

The protocol for this study served as the basis of the protocol developed by the World Health Organization (WHO) Committee on Pathobiological Determinants of Atherosclerosis in Youth. It was planned to incorporate this study into the WHO study so that cross-cultural and geographic factors could be evaluated in populations with higher and lower incidence of atherosclerosis.

DESIGN NARRATIVE:

A common protocol was followed for collecting risk factor data and coronary arteries and aortas from approximately 1,000 autopsies per year for three years. Specimens were collected and preserved in a standardized way at each collection center. Data management and statistical analysis were conducted at the University of Texas in San Antonio. The unit at Louisiana State University was composed of three central laboratories: the lipid biochemistry center; the coronary heart disease risk factor center; and a gross morphology center. The morphometry central laboratory was located at Ohio State University. Administration and coordination were directed from the University of Chicago and the University of Illinois.

In addition to serving as collection centers, many of the centers carried out individual research projects. At the University of Alabama in Birmingham, two separate but related investigations were conducted: Dr. Miller analyzed the various collagens by solubilizing them as peptide fractions and isolating the peptides via chromatography; Dr. Gay used monoclonal antibodies to define the distribution of the various collagens in atheromatous lesions. At the West Virginia University under Dr. Jagannathan, there were studies on isomeric fatty acids and proteoglycans. Dr. Reichenbach at the University of Washington studied the distribution of immunocytochemical markers of smooth muscle cell differentiation and leukocyte subpopulations in the coronary arteries as well as searched for viral DNA in plaques. At Baylor, the three-dimensional distribution of lipid inclusions, macrophages, and smooth muscle cells in coronary arteries were determined by digital fluorescence. Dr. Mergner of the University of Maryland collected specimens in the immediate autopsy program which provided specimens free of autolysis. He also performed transmission and scanning electron microscopy, X-ray microanalysis, lipid analysis, and immunofluorescence and immunoperoxidase procedures to define calcium content and cytoskeletal components. Dr. Virmani at Vanderbilt determined the role of biogenic amines such as histamine, serotonin, and catecholamines in atherosclerosis and correlated the content of amines with the presence of mast cells in the adventitia.

In 1988, two regular research grants were awarded as part of this multicenter study. The grant at the Southwest Foundation for Biomedical Research determined the genotypes for each subject with respect to restriction fragment length polymorphisms in apolipoprotein and LDL receptor genes using Southern blot analyses of DNA from liver samples sent from each collection center. It also typed the subjects for apo E isoform genotypes using oligonucleotide probes. The grant at Ohio State University correlated 3-D coronary axial geometry and pathology.

Some of the major questions addressed by the study included: whether some or all fatty streaks progressed to fibrous plaques and the transitional lesions; the morphometric and biochemical lesion changes indicated by progression; the frequency and features of insudative and proliferative lesions which may portend progressive disease; sex differences in lesions; whether immune complexes or viral infections were implicated.

In FY 1991, six grants were awarded under the title "Risk Factors in Early Human Atherogenesis" (RFEHA). The purpose was to extend the ongoing PDAY and to : obtain an adequate number of female cases so that risk factor associations could be accurately detected and studied; to increase the power of the study in general to detect associations of risk factors with raised lesions, which began to appear in this age group; and to increase the power of the study to detect genetic influences on atherosclerosis. REFHA added 1,400 new specimens to the 1,800 cases already collected in PDAY to achieve approximately 3,000 total specimens. Emphasis was placed on female cases and those that provided the best opportunity to study transition lesions between fatty streaks and fibrous plaques.

In 1998, the NHLBI awarded R24HL60808 for five years to provide and maintain an archive of human cardiovascular and other tissues which can be used by other United States and international investigators to study human atherosclerosis. The investigators, as part of PDAY and RFEHA, have assembled autopsy material (mostly of aorta and coronary artery, but with other tissues including liver, serum, and adipose tissue) from over 3,000 Black and white males and females. These were from autopsies on individuals ages 15 to 34 and obtained within 48 hours of death. The grant for the cardiovascular specimen and data library was renewed through July 2007.

ELIGIBILITY:
No eligibility criteria

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1985-06; Primary Completion 1993-07 (Actual); Study Completion 1993-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Chandler — Augusta University; J. Cornhill — Ohio State University; Asaad Daoud — Albany Medical College; Morton Friedman — Ohio State University; Steffen Gay — University of Alabama at Birmingham; James Hixson — Southwest Foundation for Biomedical Research; Singanallur Jagannathan — West Virginia University Medical Center; C. McMahan — University of Texas; Wolfgang Mergner — University of Maryland; Edward Miller — University of Alabama at Birmingham; Stanley Radio — University of Nebraska; Dennis Reichebach — University of Washington; Abel Robertson — University of Illinois at Chicago; Louis Smith — Baylor College of Medicine; Jack Strong — Louisiana State University Medical Center; Renu Virmani — Vanderbilt University School of Medicine; Robert Wissler — University of Chicago

REFERENCES:
- [Background] Relationship of atherosclerosis in young men to serum lipoprotein cholesterol concentrations and smoking. A preliminary report from the Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. JAMA. 1990 Dec 19;264(23):3018-24. doi: 10.1001/jama.1990.03450230054029. PMID 2243430
- [Background] Hixson JE, McMahan CA, McGill HC Jr, Strong JP. Apo B insertion/deletion polymorphisms are associated with atherosclerosis in young black but not young white males. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb. 1992 Sep;12(9):1023-9. doi: 10.1161/01.atv.12.9.1023. PMID 1525116
- [Background] Hixson JE. Apolipoprotein E polymorphisms affect atherosclerosis in young males. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb. 1991 Sep-Oct;11(5):1237-44. doi: 10.1161/01.atv.11.5.1237. PMID 1680392
- [Background] Wissler RW. Theories and new horizons in the pathogenesis of atherosclerosis and the mechanisms of clinical effects. Arch Pathol Lab Med. 1992 Dec;116(12):1281-91. PMID 1456873
- [Background] Wissler RW. USA Multicenter Study of the pathobiology of atherosclerosis in youth. Ann N Y Acad Sci. 1991;623:26-39. doi: 10.1111/j.1749-6632.1991.tb43716.x. No abstract available. PMID 2042833
- [Background] Wissler RW, Vesselinovitch D, Komatsu A. The contribution of studies of atherosclerotic lesions in young people to future research. Ann N Y Acad Sci. 1990;598:418-34. doi: 10.1111/j.1749-6632.1990.tb42313.x. No abstract available. PMID 2248455
- [Background] Wissler RW, Vesselinovitch D. An update on the pathogenesis of atherosclerosis (principles of prevention, intervention, retardation, and regression). Hawaii Med J. 1990 Jul;49(7):237-40, 261. PMID 2397997
- [Background] McGill HC Jr, Strong JP, Tracy RE, McMahan CA, Oalmann MC. Relation of a postmortem renal index of hypertension to atherosclerosis in youth. The Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2222-8. doi: 10.1161/01.atv.15.12.2222. PMID 7489246
- [Background] Cornhill JF, Herderick EE, Vince DG. The clinical morphology of human atherosclerotic lesions. Lessons from the PDAY Study. Pathobiological Determinants of Atherosclerosis in Youth. Wien Klin Wochenschr. 1995;107(18):540-3. PMID 7483640
- [Background] McGill HC Jr, McMahan CA, Malcom GT, Oalmann MC, Strong JP. Relation of glycohemoglobin and adiposity to atherosclerosis in youth. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb Vasc Biol. 1995 Apr;15(4):431-40. doi: 10.1161/01.atv.15.4.431. PMID 7749853
- [Background] Strong JP. Natural history and risk factors for early human atherogenesis. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Clin Chem. 1995 Jan;41(1):134-8. PMID 7813067
- [Background] Wissler RW. New insights into the pathogenesis of atherosclerosis as revealed by PDAY. Pathobiological Determinants of Atherosclerosis in Youth. Atherosclerosis. 1994 Aug;108 Suppl:S3-20. doi: 10.1016/0021-9150(94)90149-x. PMID 7802726
- [Background] Natural history of aortic and coronary atherosclerotic lesions in youth. Findings from the PDAY Study. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb. 1993 Sep;13(9):1291-8. doi: 10.1161/01.atv.13.9.1291. PMID 8364013
- [Background] Kuo CC, Grayston JT, Campbell LA, Goo YA, Wissler RW, Benditt EP. Chlamydia pneumoniae (TWAR) in coronary arteries of young adults (15-34 years old). Proc Natl Acad Sci U S A. 1995 Jul 18;92(15):6911-4. doi: 10.1073/pnas.92.15.6911. PMID 7624342
- [Background] Miller EJ, Malcom GT, McMahan CA, Strong JP. Atherosclerosis in young white males: arterial collagen and cholesterol. Matrix. 1993 Jul;13(4):289-96. doi: 10.1016/s0934-8832(11)80024-7. PMID 8412986
- [Background] Strong JP, Malcom GT, Oalmann MC. Environmental and genetic risk factors in early human atherogenesis: lessons from the PDAY study. Pathobiological Determinants of Atherosclerosis in Youth. Pathol Int. 1995 Jun;45(6):403-8. doi: 10.1111/j.1440-1827.1995.tb03476.x. PMID 7581930
- [Background] Strong JP. Atherosclerotic lesions. Natural history, risk factors, and topography. Arch Pathol Lab Med. 1992 Dec;116(12):1268-75. PMID 1456871
- [Background] Strong JP, Malcom GT, Newman WP 3rd, Oalmann MC. Early lesions of atherosclerosis in childhood and youth: natural history and risk factors. J Am Coll Nutr. 1992 Jun;11 Suppl:51S-54S. doi: 10.1080/07315724.1992.10737984. PMID 1619200
- [Background] Scanlon CE, Berger B, Malcom G, Wissler RW. Evidence for more extensive deposits of epitopes of oxidized low density lipoprotein in aortas of young people with elevated serum thiocyanate levels. PDAY Research Group. Atherosclerosis. 1996 Mar;121(1):23-33. doi: 10.1016/0021-9150(95)05672-6. PMID 8678921
- [Background] Botti TP, Amin H, Hiltscher L, Wissler RW. A comparison of the quantitation of macrophage foam cell populations and the extent of apolipoprotein E deposition in developing atherosclerotic lesions in young people: high and low serum thiocyanate groups as an indication of smoking. PDAY Research Group. Pathobiological Determinants of Atherosclerosis in Youth. Atherosclerosis. 1996 Aug 2;124(2):191-202. doi: 10.1016/0021-9150(96)05825-x. PMID 8830932
- [Background] Komatsu A, Sakurai I. A study of the development of atherosclerosis in childhood and young adults: risk factors and the prevention of progression in Japan and the USA. The Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Pathol Int. 1996 Aug;46(8):541-7. doi: 10.1111/j.1440-1827.1996.tb03652.x. PMID 8893222
- [Background] Wissler RW, Group PD. Atheroarteritis: a combined immunological and lipid imbalance. Int J Cardiol. 1996 Aug;54 Suppl:S37-49. doi: 10.1016/s0167-5273(96)88772-9. PMID 9119526
- [Background] Strong JP, Malcom GT, Oalmann MC, Wissler RW. The PDAY Study: natural history, risk factors, and pathobiology. Pathobiological Determinants of Atherosclerosis in Youth. Ann N Y Acad Sci. 1997 Apr 15;811:226-35; discussion 235-7. doi: 10.1111/j.1749-6632.1997.tb52004.x. No abstract available. PMID 9186600
- [Background] Malcom GT, Oalmann MC, Strong JP. Risk factors for atherosclerosis in young subjects: the PDAY Study. Pathobiological Determinants of Atherosclerosis in Youth. Ann N Y Acad Sci. 1997 May 28;817:179-88. doi: 10.1111/j.1749-6632.1997.tb48205.x. No abstract available. PMID 9239187
- [Background] Kuhn H, Heydeck D, Hugou I, Gniwotta C. In vivo action of 15-lipoxygenase in early stages of human atherogenesis. J Clin Invest. 1997 Mar 1;99(5):888-93. doi: 10.1172/JCI119253. PMID 9062346
- [Background] McGill HC Jr, McMahan CA, Malcom GT, Oalmann MC, Strong JP. Effects of serum lipoproteins and smoking on atherosclerosis in young men and women. The PDAY Research Group. Pathobiological Determinants of Atherosclerosis in Youth. Arterioscler Thromb Vasc Biol. 1997 Jan;17(1):95-106. doi: 10.1161/01.atv.17.1.95. PMID 9012643
- [Background] Zieske AW, Takei H, Fallon KB, Strong JP. Smoking and atherosclerosis in youth. Atherosclerosis. 1999 Jun;144(2):403-8. doi: 10.1016/s0021-9150(98)00326-8. PMID 10407501
- [Background] Rainwater DL, McMahan CA, Malcom GT, Scheer WD, Roheim PS, McGill HC Jr, Strong JP. Lipid and apolipoprotein predictors of atherosclerosis in youth: apolipoprotein concentrations do not materially improve prediction of arterial lesions in PDAY subjects. The PDAY Research Group. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):753-61. doi: 10.1161/01.atv.19.3.753. PMID 10073983
- [Background] McGill HC Jr, McMahan CA, Tracy RE, Oalmann MC, Cornhill JF, Herderick EE, Strong JP. Relation of a postmortem renal index of hypertension to atherosclerosis and coronary artery size in young men and women. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb Vasc Biol. 1998 Jul;18(7):1108-18. doi: 10.1161/01.atv.18.7.1108. PMID 9672071
- [Background] McGill HC Jr, McMahan CA. Determinants of atherosclerosis in the young. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Am J Cardiol. 1998 Nov 26;82(10B):30T-36T. doi: 10.1016/s0002-9149(98)00720-6. PMID 9860371
- [Background] Wissler RW, Strong JP. Risk factors and progression of atherosclerosis in youth. PDAY Research Group. Pathological Determinants of Atherosclerosis in Youth. Am J Pathol. 1998 Oct;153(4):1023-33. doi: 10.1016/s0002-9440(10)65647-7. No abstract available. PMID 9777934
- [Background] Strong JP, Malcom GT, McMahan CA, Tracy RE, Newman WP 3rd, Herderick EE, Cornhill JF. Prevalence and extent of atherosclerosis in adolescents and young adults: implications for prevention from the Pathobiological Determinants of Atherosclerosis in Youth Study. JAMA. 1999 Feb 24;281(8):727-35. doi: 10.1001/jama.281.8.727. PMID 10052443
- [Background] Sloop GD, Perret RS, Brahney JS, Oalmann M. A description of two morphologic patterns of aortic fatty streaks, and a hypothesis of their pathogenesis. Atherosclerosis. 1998 Nov;141(1):153-60. doi: 10.1016/s0021-9150(98)00167-1. PMID 9863548
- [Background] Wissler RW. An overview of the quantitative influence of several risk factors on progression of atherosclerosis in young people in the United States. Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Am J Med Sci. 1995 Dec;310 Suppl 1:S29-36. doi: 10.1097/00000441-199512000-00006. PMID 7503120
- [Background] McGill HC Jr, McMahan CA, Zieske AW, Tracy RE, Malcom GT, Herderick EE, Strong JP. Association of Coronary Heart Disease Risk Factors with microscopic qualities of coronary atherosclerosis in youth. Circulation. 2000 Jul 25;102(4):374-9. doi: 10.1161/01.cir.102.4.374. PMID 10908207
- [Background] McGill HC Jr, McMahan CA, Herderick EE, Tracy RE, Malcom GT, Zieske AW, Strong JP. Effects of coronary heart disease risk factors on atherosclerosis of selected regions of the aorta and right coronary artery. PDAY Research Group. Pathobiological Determinants of Atherosclerosis in Youth. Arterioscler Thromb Vasc Biol. 2000 Mar;20(3):836-45. doi: 10.1161/01.atv.20.3.836. PMID 10712411
- [Background] Zieske AW, Malcom GT, Strong JP. Pathobiological determinants of atherosclerosis in youth (PDAY) cardiovascular specimen and data library. J La State Med Soc. 2000 Jun;152(6):296-301. PMID 10935370
- [Background] McGill HC Jr, McMahan CA, Zieske AW, Malcom GT, Tracy RE, Strong JP. Effects of nonlipid risk factors on atherosclerosis in youth with a favorable lipoprotein profile. Circulation. 2001 Mar 20;103(11):1546-50. doi: 10.1161/01.cir.103.11.1546. PMID 11257083
- [Background] McGill HC Jr, McMahan CA, Zieske AW, Sloop GD, Walcott JV, Troxclair DA, Malcom GT, Tracy RE, Oalmann MC, Strong JP. Associations of coronary heart disease risk factors with the intermediate lesion of atherosclerosis in youth. The Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Arterioscler Thromb Vasc Biol. 2000 Aug;20(8):1998-2004. doi: 10.1161/01.atv.20.8.1998. PMID 10938023
- [Background] Rao RN, Falls DG, Gerrity RG, Sethuraman SN, Thiruvaiyaru DS. Intimal thickness and layering, and smooth muscle cell phenotypes in aorta of youth. Pathobiology. 2000 Jan-Feb;68(1):18-28. doi: 10.1159/000028111. PMID 10859527
- [Background] Zieske AW, Malcom GT, Strong JP. Natural history and risk factors of atherosclerosis in children and youth: the PDAY study. Pediatr Pathol Mol Med. 2002 Mar-Apr;21(2):213-37. doi: 10.1080/15227950252852104. PMID 11942537
- [Background] Millonig G, Malcom GT, Wick G. Early inflammatory-immunological lesions in juvenile atherosclerosis from the Pathobiological Determinants of Atherosclerosis in Youth (PDAY)-study. Atherosclerosis. 2002 Feb;160(2):441-8. doi: 10.1016/s0021-9150(01)00596-2. PMID 11849669
- [Background] Ishikawa Y, Ishii T, Akasaka Y, Masuda T, Strong JP, Zieske AW, Takei H, Malcom GT, Taniyama M, Choi-Miura NH, Tomita M. Immunolocalization of apolipoproteins in aortic atherosclerosis in American youths and young adults: findings from the PDAY study. Atherosclerosis. 2001 Sep;158(1):215-25. doi: 10.1016/s0021-9150(01)00416-6. PMID 11500194
- [Background] Homma S, Ishii T, Malcom GT, Zieske AW, Strong JP, Tsugane S, Hirose N. Histopathological modifications of early atherosclerotic lesions by risk factors--findings in PDAY subjects. Atherosclerosis. 2001 Jun;156(2):389-99. doi: 10.1016/s0021-9150(00)00669-9. PMID 11395036
- [Background] McGill HC Jr, McMahan CA, Herderick EE, Zieske AW, Malcom GT, Tracy RE, Strong JP; Pathobiological Determinants of Atherosclerosis in Youth (PDAY) Research Group. Obesity accelerates the progression of coronary atherosclerosis in young men. Circulation. 2002 Jun 11;105(23):2712-8. doi: 10.1161/01.cir.0000018121.67607.ce. PMID 12057983
- [Background] McGill HC Jr, Herderick EE, McMahan CA, Zieske AW, Malcolm GT, Tracy RE, Strong JP. Atherosclerosis in youth. Minerva Pediatr. 2002 Oct;54(5):437-47. PMID 12244281
- [Background] Strong JP, Zieske AW, Malcom GT. Lipoproteins and atherosclerosis in children: an early marriage? Nutr Metab Cardiovasc Dis. 2001 Oct;11 Suppl 5:16-22. PMID 12063771
- [Background] Cohen HW, Sloop GD; PDAY Study. Glucose interaction magnifies atherosclerotic risk from cholesterol. Findings from the PDAY Study. Atherosclerosis. 2004 Jan;172(1):115-20. doi: 10.1016/j.atherosclerosis.2003.09.010. PMID 14709364
- [Background] McMahan CA, Gidding SS, Fayad ZA, Zieske AW, Malcom GT, Tracy RE, Strong JP, McGill HC Jr. Risk scores predict atherosclerotic lesions in young people. Arch Intern Med. 2005 Apr 25;165(8):883-90. doi: 10.1001/archinte.165.8.883. PMID 15851639
- [Background] Zieske AW, McMahan CA, McGill HC Jr, Homma S, Takei H, Malcom GT, Tracy RE, Strong JP. Smoking is associated with advanced coronary atherosclerosis in youth. Atherosclerosis. 2005 May;180(1):87-92. doi: 10.1016/j.atherosclerosis.2004.10.039. Epub 2004 Dec 15. PMID 15823279
- [Background] Scheer WD, Boudreau DA, Hixson JE, McGill HC, Newman WP 3rd, Tracy RE, Zieske AW, Strong JP. ACE insert/delete polymorphism and atherosclerosis. Atherosclerosis. 2005 Feb;178(2):241-7. doi: 10.1016/j.atherosclerosis.2004.09.019. PMID 15694930
- [Background] Wissler RW. Update on the pathogenesis of atherosclerosis. Am J Med. 1991 Jul 31;91(1B):3S-9S. doi: 10.1016/0002-9343(91)90050-8. PMID 1867233